CLINICAL TRIAL: NCT04876313
Title: An Open Label, Single-arm, Phase 2 Study of Neoadjuvant Nivolumab and Nab-paclitaxel Before Radical Cystectomy for Patients With Muscle-invasive Bladder Cancer
Brief Title: An Open Label, Single-arm, Phase 2 Study of Neoadjuvant Nivolumab and Nab-paclitaxel Before Radical Cystectomy for Patients With Muscle-invasive Bladder Cancer (NURE-Combo)
Acronym: NURE-Combo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Prof. Andrea Necchi, Associate Professor - Head of Genitourinary Medical Oncology, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NURE-Combo; 2020-005050-20 (EudraCT Number)
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Muscle-Invasive Bladder Carcinoma
MeSH Terms: interventions — Nivolumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Patients with muscle-invasive urothelial bladder carcinoma, not eligible or denying standard neoadjuvant therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Drugs (Experimental): Participants received 4x3 weekly cycles of 360 mg Nivolumab + 125 mg/m^2 Nab-paclitaxel IV on days 1 and 8, then they had cystectomy after that partecipants received adjuvant nivolumab 360 mg IV Q3W X13 cycles
  Interventions: Drug: Nivolumab + Nab-paclitaxel; Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab + Nab-paclitaxel — 4x3 weekly cycles of 360 mg nivolumab + 125 mg/m^2 nab-paclitaxel IV on days 1 and 8
  Other Names: Nivolumab + Abraxane
Drug: Nivolumab — 360 mg IV Q3W x 13 cycles
  Other Names: Adjuvant Nivolumab

SUMMARY:
To assess whether nivolumab+nab-paclitaxel combination results in patients with muscle-invasive bladder cancer

DETAILED DESCRIPTION:
This is a Phase 2, single-center, open-label, non-randomized study in patients with muscle-invasive urothelial carcinoma of the bladder.

The general framework of the study will be as follows:

A transurethral resection of the bladder for biopsy, histological characterization, and local staging will be executed first. With the aim to improve the sensitivity of CT scan in assessing pelvic lymph-nodes and better assess the local extent of bladder tumor, computed tomography (CT) scan, 18FDG-PET/CT scan, and multiparametric bladder MRI (mpMRI) will be done during screening and before cystectomy to stage and evaluate response.

Eligible patients will receive neoadjuvant treatment: 360 mg nivolumab IV on Day 1 plus 125 mg/m2 nab-paclitaxel on Day 1 and 8, in a 21-day cycle.

A total of 4 cycles are planned before surgery. Surgery will be planned at the time of study inclusion to be done within 3 weeks of the last dose of study drug.

Dose reductions will be applied depending on the severity of AEs, and treatment interruption or discontinuation criteria will be fully described in the protocol.

After surgery, patients will receive 12-month adjuvant therapy with nivolumab 360 mg IV, every 3 weeks.

RECIST v1.1 criteria will be used to assess patient response to treatment by determining tumor size and PFS. Screening assessments should be performed no more than 21 days prior to the start of study treatment. Following the screening assessment, subsequent assessments will be carried out after the administration of the study drugs prior to cystectomy. If an unscheduled assessment is performed and the patient has not progressed, the results should be reported at the next scheduled visit. The method of tumor assessment used at baseline e.g. CT or MRI scans chest, abdomen, pelvis, must be used at each sub-sequent follow-up assessment.

Patients will be monitored carefully for the development of adverse events and will be monitored for clinical and/or radiographic evidence of disease progression according to usual standards of clinical practice. Adverse experiences will be evaluated according to criteria outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects, >18 years of age, able to understand and give written informed consent.
* Histopathologically confirmed urothelial carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) transitional cell pattern.
* Fit and planned for RC (according to local guidelines).
* ECOG performance status score of 0 or 1.
* Adequate hematologic counts without transfusional or growth factor support within 2 weeks of study drug initiation (Hemoglobin ≥ 9 g/dL, ANC ≥ 1,500/ mm3, and Platelets ≥ 100,000/ μL).
* Adequate hepatic function (Bilirubin ≤ 1.5 IULN, AST and ALT ≤ 2.5 x IULN or ≤ 5 x IULN if known liver metastases and serum albumin >3 g/dl).
* Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication, and must not be lactating. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 4 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >2 years.
* Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy.
* Clinical stage T2-T4aN0M0 MIBC, assessed by CT + PET/CT + mpMRI.
* The patient accepts to undergo RC.
* Ineligibility to receive cisplatin-based neoadjuvant chemotherapy based on Galsky's criteria (Galsky MD, et al. J Clin Oncol. 2011 Jun 10;29(17):2432-8) OR refusal to receive neoadjuvant cisplatin-based chemotherapy.

Exclusion Criteria:

* Has received prior systemic anti-cancer therapy including investigational agents and immunotherapy.
* Prior immunotherapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137.
* Has received prior radiotherapy on the bladder tumor.
* Have received a partial cystectomy.
* Refusal to undergo RC.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has received any antibiotics within 30 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Participants with low-risk early stage prostate cancer defined as follows are not excluded; Stage T1c or T2a with a Gleason score ≤ 6 and prostatic-specific antigen (PSA) < 10 ng/mL either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to study allocation.
* Has severe hypersensitivity (≥Grade 3) to nivolumab or nab-paclitaxel and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Have active cardiac disease, defined as:

  * Myocardial infarction or unstable angina pectoris within 6 months of C1D1
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation
  * NYHA Class III or greater congestive heart failure or left ventricular ejection fraction of < 40%
* Have known history of HIV-1/2 infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Have other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* High dose systemic corticosteroids (≥20 mg of prednisolone or its equivalent) are not allowed within 2 weeks of C1D1.
* Have received or are currently receiving (within the previous 2 weeks) antibiotics.
* Have a pre-existing motor or sensory neuropathy of a severity >= grade 2 by NCI-CTC criteria due to the potential for neuropathy of nab-paclitaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Change from Screening after radical cystectomy
  To assess whether nab-paclitaxel plus nivolumab results in pathological complete response (herein referred to as either "ypT0N0M0" or "pCR") in patients with clinical T2-4aN0M0 MIBC who cannot receive or refuse to receive cisplatin-based chemotherapy. Absence of any residual viable tumor in the radical cystectomy specimen. Two independent pathologists, blinded to the study findings, with >10 years of experience in genitourinary tumors will independently evaluate the response.

SECONDARY OUTCOMES:
pathological downstaging | screening, 14 days after final combined treatment, 3 weeks until 12 months post-radical cystectomy, 3 months until 12 months post-adjuvant nivolumab
  To evaluate the proportion of patients who will be pathological downstaged to ypT<=1N0M0.
radiological response | screening, 14 days after final combined treatment, 3 weeks until 12 months post-radical cystectomy, 3 months until 12 months post-adjuvant nivolumab
  To evaluate radiological response on those patients with measurable disease. Response (CR and PR) will be assessed after the full neoadjuvant course of 4 cycles.
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 and EAU recommendations | From date of Screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  To evaluate the surgical and medical safety of neoadjuvant combination therapy, as well as of the adjuvant nivolumab therapy.
event-free survival | From date of Screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  To assess event-free survival in the total population and in the subgroups according to the pathological response.
overall survival | From date of Screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  To assess overall survival in the total population and in the subgroups according to the pathological response.

CONTACTS AND LOCATIONS:
Locations (1):
- Genitourinary Medical Oncology - IRCCS San Raffaele Hospital and Scientific Institute, Milan, MI, Italy

REFERENCES:
- [Derived] Mercinelli C, Moschini M, Cigliola A, Mattorre B, Tateo V, Basile G, Cogrossi LL, Maiorano BA, Patane DA, Raggi D, Pastorino GL, Re C, Colecchia M, Luciano R, Colombo R, Brembilla G, De Cobelli F, Briganti A, Pavlick DC, Ross JS, Montorsi F, Bellone M, Necchi A. First Results of NURE-Combo: A Phase II Study of Neoadjuvant Nivolumab and Nab-Paclitaxel, Followed by Postsurgical Adjuvant Nivolumab, for Muscle-Invasive Bladder Cancer. J Clin Oncol. 2024 Dec 10;42(35):4196-4205. doi: 10.1200/JCO.24.00576. Epub 2024 Sep 6. PMID 39241203